CLINICAL TRIAL: NCT04931602
Title: Determining Feasibility of a Model of Care for Secondary Fracture Prevention for Implementation in Health Care System in Pakistan After Hip Fracture: a Clinical Outcome Study
Brief Title: Determining Feasibility of a Model of Care for Secondary Fracture Prevention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sibtain Ahmed, Assistant Professor, Aga Khan University
Other Study IDs: 2020-3409-14191
Record Dates: First submitted 2021-06-09; First posted 2021-06-18 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Osteoporosis
Keywords: Hip fractures; fracture; prevention
MeSH Terms: conditions — Osteoporosis; Hip Fractures; Fractures, Bone | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Model A: Patients will be followed-up at bone, endocrine and rheumatology clinic after discharge depending upon availability of the consultant. Multifaceted risk-factor assessment for identifying patients at risk will be conducted including formal future fracture risk assessment/life style/medication review and fall risk assessment.
  Comprehensive laboratory designed package including calcium (Ca), albumin (ALB), phosphate (P), bone alkaline phosphatase (BAP), C terminal peptide of type 1 collagen (CTx), vitamin D (25OHD) and intact parathyroid hormone (iPTH) will be performed at first clinic visit for all patients between 6-8 weeks post fracture. Screening for secondary causes of osteoporosis will be conducted for those identified in need. BMD testing as per guidelines for patients with fragility fractures will be conducted at clinic visit and recorded with risk assessment form (12).
  Interventions: Diagnostic Test: Biochemical markers i.e. Serum Ca, PTH, CTX, Albumin, Phosphate, Vitamin D and Bone mineral density Scan
- Model B: All routine intervention except treatment initiation-the responsibility of patient's general practitioner for prevention of secondary fracture. Those included in this intervention arm, will be identified and risk assessment will be performed at hospital admission. Recommendations for the treatment will be made to be initiated by the patient's general physician. Patients will be followed at 6 months on telephone, and a questionnaire related to treatment compliance &/or non-compliance will be filled by the coordinator.
  Interventions: Diagnostic Test: Biochemical markers i.e. Serum Ca, PTH, CTX, Albumin, Phosphate, Vitamin D and Bone mineral density Scan
- Model C: Health education only provided at the time of admission with handover to family physician for follow-up. Patients will be given an appointment to follow-up at community health center of Aga Khan University
  Interventions: Diagnostic Test: Biochemical markers i.e. Serum Ca, PTH, CTX, Albumin, Phosphate, Vitamin D and Bone mineral density Scan
- Model D: Health Education provided. There is no physician contact with the person's general practitioner for prevention of secondary fracture. Education material for the patient have been prepared and will be provided to patient along with counselling by the nurse at the time of discharge
  Interventions: Diagnostic Test: Biochemical markers i.e. Serum Ca, PTH, CTX, Albumin, Phosphate, Vitamin D and Bone mineral density Scan

INTERVENTIONS:
Diagnostic Test: Biochemical markers i.e. Serum Ca, PTH, CTX, Albumin, Phosphate, Vitamin D and Bone mineral density Scan — investigations for secondary causes of osteoporosis

SUMMARY:
Osteoporosis is a disorder of low bone mass and micro-architectural deterioration resulting in decreased mechanical strength and increased susceptibility to fractures even after minimal trauma. These 'minimal trauma fractures' (also known as 'osteoporotic', 'low trauma' or 'fragility' fractures) are the hallmark of a chronic and disabling disease that affects both men and women worldwide. On statistical grounds, more than 50 % of postmenopausal women and 30 % of men over the age of 60 years will suffer at least one minimal trauma fracture during their remaining lifetime. Any osteoporotic fracture predisposes to further fractures, significant morbidity and premature death. Thus, following a first minimal trauma fracture both men and women have a two- to threefold increased risk of subsequent fracture.

This study aims to determine feasibility of evaluating different models of care through a structured multidisciplinary path tailored to identify, assess and treat hip fracture patients in an effective timely manner that are at high risk of subsequent fracture (Type A model) and to compare its effectiveness and feasibility with a type B, C & D model as proposed by Ganda et al at the Aga Khan University, with collaboration of the departments of Orthopaedics, Chemical Pathology, Family Medicine and Internal Medicine.

DETAILED DESCRIPTION:
With the severity of implications associated with fragility fractures, prevention of a secondary fracture has become a primary focus from a patient care and societal standpoint worldwide. However, this area has been so far neglected in Pakistan. A fracture requires that two conditions occur simultaneously: week bones and a fall or stress on week bones and a co-management approach is required to address both issues.

The investigators propose to determine feasibility of evaluating different models of care through a structured multidisciplinary path tailored to identify, assess and treat hip fracture patients in an effective timely manner that are at high risk of subsequent fracture (Type A model) and to compare its effectiveness and feasibility with a type B, C & D model as proposed by Ganda et al. Based on this study the investigators will propose a model of care for SFP for application at national level in private and public sector. The long-term plan is to develop a national fragility fracture network in preventing and managing fragility fractures and to promote research aimed at better treatments of osteoporosis, sarcopenia and fracture in line with global CtA from FFN. This information will also help us in applying clinical practice guidelines for osteoporosis and driving policy change for our country which is currently non-existent and is likely to be a step towards the achievement of Sustainable Development Goals (SDG) (i.e. ensure healthy lives and promote wellbeing for all at all ages) and in line with WHO decade of healthy ageing 2021-23.

Specific Aims:

This study is primarily aimed at comparison of the feasibility and effectiveness of models of care (Type A, B, C & D) for hip fracture patients. The Specific, Measurable, Achievable, Realistic, and Time-defined (SMART) goals of this project are formulated around the 5IQ approach delineated by the Royal Osteoporosis society based on the following 6 parameters.

I. Identification: systematic screening of high-risk individuals

II. Investigation: undertaking of relevant investigations to delineate the cause of low bone mass

III. Information: educating patients on falls prevention and fracture risk

IV. Initiation: provision of pharmacological, lifestyle, dietary, conservative management approach and falls prevention interventions according to the model of care adopted

V. Integration: promotion of integration between primary and secondary care

VI. Quality: Ensuring professional development, audit, and peer-review activities

Type A model: Intensive service with all routine interventions:

Participants will be followed-up at bone, endocrine and rheumatology clinic after discharge depending upon availability of the consultant. Multifaceted risk-factor assessment for identifying patients at risk will be conducted including formal future fracture risk assessment/life style/medication review and fall risk assessment.

Comprehensive laboratory designed package including calcium (Ca), albumin (ALB), phosphate (P), bone alkaline phosphatase (BAP), C terminal peptide of type 1 collagen (CTx), vitamin D (25OHD) and intact parathyroid hormone (iPTH) will be performed at first clinic visit for all patients between 6-8 weeks post fracture. Screening for secondary causes of osteoporosis will be conducted for those identified in need. BMD testing as per guidelines for patients with fragility fractures will be conducted at clinic visit and recorded with risk assessment form.

Type B model: All intervention except treatment initiation-the responsibility of participants general practitioner for prevention of secondary fracture Those included in this intervention arm, will be identified and risk assessment will be performed at hospital admission. Recommendations for the treatment will be made to be initiated by the patient's general physician. Participants will be followed at 6 months on telephone, and a questionnaire related to treatment compliance &/or non-compliance will be filled by the coordinator.

Type C model: Health education only provided at the time of admission with handover to family physician for follow-up. Participants will be given an appointment to follow-up at community health center of Aga Khan University.

Type D model: Health Education provided. There is no physician contact with the participant's general practitioner for prevention of secondary fracture. Education material for the patient have been prepared and will be provided to the participant along with counselling by the nurse at the time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* All women ≥50 years with low trauma hip fracture
* All post-menopausal women ( less than 50 years) with low trauma hip fracture
* Men ≥50 years with low trauma hip fracture

Exclusion Criteria:

• Patients with high impact hip fracture including after road traffic accident

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with low trauma hip fractures at the out-patients or at emergency department
Sampling Method: Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Secondary fracture prevention of hip | 1 year of follow-up
  Rate of Secondary fracture of hip (occurrence of hip fracture (n) if any during the follow up will be noted)
Total Secondary fracture prevention | 1 year of follow-up
  Rate of total fracture (occurrence of fracture (n), if any, during the follow up will be noted)

SECONDARY OUTCOMES:
Effectiveness of the models of care- Follow up plan | 1 year of follow-up
  On a Likert's scale of 1 to 5, rating will be recorded from the participants for: The plan for follow-up was explained to the participant clearly
Effectiveness of the models of care- Care provided post fracture | 1 year of follow-up
  On a Likert's scale of 1 to 5, rating will be recorded from the participants for: Participant is satisfied with the care provided post fracture.
Effectiveness of the models of care- Adequacy of information provided | 1 year of follow-up
  On a Likert's scale of 1 to 5, rating will be recorded from the participants for: right amount of information was given to the participant for secondary fracture prevention
Effectiveness of the models of care- Communication | 1 year of follow-up
  On a Likert's scale of 1 to 5, rating will be recorded from the participants for: The plan for managements for secondary fracture prevention was communicated adequately

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No